CLINICAL TRIAL: NCT06520956
Title: Improving Healthy Lifestyle Behaviors and Quality of Life of Elderly Individuals Living in Nursing Homes by Increasing Their Physical Activity Levels
Brief Title: Improving the Quality of Life of Elderly Individuals Living in Nursing Homes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Galata University (Other)
Responsible Party: Principal Investigator, Safak Yigit, PhD(c), Istanbul Galata University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GalataU
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Elderly People
Keywords: Brain Breaks® (BB) videos; physical activity; quality of life; walking; health lifestyle
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-based exercise group (Experimental): In each session, 2 videos will be applied and each will be repeated 2-3 times, with a 3-minute rest break between each video. The total session will last an average of 20-30 minutes and 16 sessions of physical activity will be performed twice a week for a total of 8 weeks. A total of at least 140 GCH Brain Breaks® videos, each 3-4 minutes long, include aerobic exercises that include large joint movements, yoga and movements specific to different sports branches such as volleyball, basketball, football, tennis, karate, judo, warm-up and cool-down movements. includes national dances of different cultures
  Interventions: Behavioral: Video based exercise group
- Control group (No Intervention): Any intervention will not be performed. After the initial evaluation, patients in this group will be given a single session of training on balance and posture exercises.

INTERVENTIONS:
Behavioral: Video based exercise group — In each session, 2 videos will be applied and each will be repeated 2-3 times, with a 3-minute rest break between each video. The total session will last an average of 20-30 minutes and 16 sessions of physical activity will be performed twice a week for a total of 8 weeks.
  Arms: Video-based exercise group

SUMMARY:
The development of physical activity (PA) and exercise habits improves strength, flexibility, balance and coordination, activities such as walking, sleep quality and cognitive status in elderly people and supports their participation in social life. The aim of the study is to examine the effects of web-based Brain Breaks® (BB) video exercises (study group-WG) and posture and balance exercises (control group-CG) on the general physical condition, sleep quality and life satisfaction of elderly individuals. We expect this situation to improve the healthy lifestyle behaviors of elderly individuals.

This study, planned to be conducted in two nursing homes, was planned as Evaluation-BB Physical Activity/Posture and Balance Exercises-Evaluation-1 month follow-up. Participants' sociodemographic characteristics, blood pressure, pulse, respiration, height, weight, muscle strength and flexibility, walking performance, posture, sleep and quality of life and life satisfaction will be evaluated. After the first evaluation, 2-3 BB video exercises will be applied to the study group (total n = 140 videos, t = 3-4 min) and posture and balance exercises (t = 20 min) to the control group, two days a week for 8 weeks, for a total of 16 sessions. During the follow-up period, physical activity habits will be questioned through weekly telephone calls (n = 4). All statistical analyzes will be performed in SPSS 26.0 program, and p value <0.05 will be considered statistically significant. Differences within and between groups and relationships between data and factors affecting these data will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years or older,
* There is no health problem determined by the doctor that prevents physical activity,
* Volunteering to participate in the study.

Exclusion Criteria:

* Having a serious life-threatening chronic disease or dementia,
* Having chronic or acute pain that prevents you from continuing to work,
* Having uncontrolled hypotension/hypertension, cardiovascular problems, metabolic and chronic diseases

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Six Minute Walking Test | At baseline and at week 8
  It is a test used to evaluate an individual's aerobic capacity. Individuals are asked to walk as much as possible for 6 minutes in a corridor that is at least 30 meters long and has a flat and hard surface. The distance traveled in 6 minutes is recorded. While the average walking distance is 570 meters for men aged 50-70 and 540 meters for women; It is stated as 530 meters for men aged 70-80 and 470 meters for women. Test results lower than these values may be associated with a decrease in aerobic capacity (American Thoracic Society 2002).

SECONDARY OUTCOMES:
Posture Evaluation | At baseline and at week 8
  People's postures were evaluated with the New York Posture Assessment Test on thirteen (13) parts of the body from the back (head-A, shoulder levels-B, vertebral column-C, hip levels-D, mediolateral position of the feet-E, foot arches-F) and side ( head-G, rib cage-H, shoulders-I, upper back-J, trunk-K, abdomen-L, lower back-waist-M) will be observed and scored on the form. Accordingly, five (5) points will be given if the posture of the examined area is good, three (3) points will be given if it is moderately damaged, and one (1) point will be given if it is seriously damaged. The total score obtained as a result of the test is a maximum of 65 and a minimum of 13. Accordingly, if the score is 45, it will be classified as 'very good', if it is between 40-44, it will be classified as 'good', if it is 30-39, it will be classified as 'medium', if it is 20-29, it will be classified as poor and if it is 19, it will be classified as 'bad'.
Healthy Lifestyle Behaviors Scale II | At baseline and at week 8
  The Healthy Lifestyle Behaviors Scale, developed by Walker et al. (1987), was revised in 1996 and named Healthy Lifestyle Behaviors Scale II. The alpha value of the scale, which has a total of 52 items and 6 sub-factors (health responsibility, physical activity, nutrition, spiritual development, interpersonal relations, stress management), was determined as 0.94. A high total score indicates that there are more healthy lifestyle behaviors (Bahar et al., 2008).
Sleep quality | At baseline and at week 8
  Sleep quality will be evaluated with the Pittsburg Sleep Quality Index (PSQI), developed by Buysse et al. (1989) and adapted into Turkish by Ağargün et al. (1996). PSQI is a 19-item self-report scale that evaluates sleep quality and disturbance over the past month. It consists of 24 questions. 19 questions are self-report questions, 5 questions are questions to be answered by the spouse or roommate. The 18 scored questions of the scale consist of 7 components: Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disturbance, Sleeping Medication Use, and Daytime Dysfunction. Each component is evaluated on a scale of 0-3 points. The total score of the 7 components gives the total score of the scale. Total score varies between 0-21. A total score greater than 5 indicates "poor sleep quality".
Life Satisfaction Scale | At baseline and at week 8
  To evaluate life satisfaction, the Content with Life Scale, consisting of 5 items developed by Lavallee et al. (2007), will be used (27). This one-dimensional scale has a 7-point Likert-type rating ("1" strongly disagree - "7" strongly agree). Turkish validity and reliability analysis was conducted by Akın and Yalnız (2015), and high scores indicate a high level of life satisfaction.
Flexibility assessment | At baseline and at week 8
  For Shortness-Flexibility evaluation, shoulder (Apley test) and lower extremity flexibility (sit-reach test) (short:3, moderately short:2 and normal:1) will be tested. Measurements will be taken separately for the right and left side of the body.
Barthel Index | At baseline and at week 8
  The index developed by Mahoney and Barthel in 1965 was modified by Shah et al. (1992). This scale evaluates mobility status and stair climbing functions such as feeding, washing, self-care, dressing, defecation control, urinary control, going to the toilet, ability to move from bed to wheelchair, walking or being dependent on a wheelchair, and stair climbing on a scale of 5-15 points (depending on the question). It consists of a total of 10 items that grade each other (0-15 points in 5-point increments).

CONTACTS AND LOCATIONS:
Overall Officials: Habibe Serap Inal, Prof.Dr., Study Director — Istanbul Galata University; Gülenay Yıldırım, MsC, Principal Investigator — Istanbul Galata University; Büşra Ülker Ekşi, PhD(c), Study Chair — Istanbul Galata University; Şafak Yiğit, PhD(c), Study Chair — Istanbul Galata University; Nejla Uzun, PhD, Study Chair — Istanbul Galata University; Alihan Bilen, PhD(c), Study Chair — Istanbul Galata University
Locations (1):
- Istanbul Galata University, Istanbul, Beyoğlu, Turkey (Türkiye)